CLINICAL TRIAL: NCT05884138
Title: A Randomized Controlled Trial to Analyze the Effects of Essential Aminoacid Supplementation and Exercise on the Improvement of Skeletal Muscle Function in Hemodialysis Patients
Brief Title: Effect of Essential Aminoacid Supplementation and Exercise on Skeletal Muscle Function in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-ED-2023-001
Record Dates: First submitted 2023-05-18; First posted 2023-06-01 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenia
Keywords: hemodialysis; nutrition; exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Exercise; Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Improved skeletal muscle function due to protein supplementation and exercise (Experimental): resistance exercise and protein supplementation including branched chain amino acids for 12 weeks
  Interventions: Other: exercise and nutritional support
- control (No Intervention): No intervention, but the same measurements as the experimental group are conducted.

INTERVENTIONS:
Other: exercise and nutritional support — resistance exercise and protein supplementation including branched chain amino acids for 12 weeks
  Arms: Improved skeletal muscle function due to protein supplementation and exercise

SUMMARY:
Sarcopenia can be easily observed in patients with hemodialysis. However, there were few studies on the precise concept and diagnostic criteria for sarcopenia in patients with hemodialysis. The investigators have already recognized the sarcopenia-associated mortality and morbidity in patients with hemodialysis. However, intervention studies on hemodialysis patients with sarcopenia have not been conducted until now. In 2021, the investigators conducted a pilot study to evaluate the effectiveness of the combined exercise and nutrition intervention for sarcopenia in patients with hemodialysis to confirm the effectiveness. This study is a follow-up study, conducted as a randomized controlled trial.

DETAILED DESCRIPTION:
This is a prospective, 1:1 randomized controlled study with 40 patients with hemodialysis who were diagnosed as sarcopenia or frailty in our previous cohort study. Combined intervention will consist of resistance exercise and nutritional supplementation for 12 weeks. The primary outcome of this study is muscle mass and handgrip strength after 12 weeks' intervention. All functional outcomes will be measured at 0, 4, 8 and 12 weeks after intervention. The data will be analysed using the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemodialysis
* Community-dwellers
* Able to walk with or without assistive devices for more than 100 meters

Exclusion Criteria:

* A person with cancer disease.
* People with psychiatric symptoms.
* A person who has an absorption disorder or has a history of resection of the small intestine or colon
* Pregnant women
* A person treated for acute bacterial infections
* A person who is in a wheelchair due to inconvenience in walking.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength in Kg using a portable dyanometer | 12 weeks
  Measurement of handle strength using a portable dynamometer to view the function of skeletal muscle every 4 weeks.
Body composition using dual energy x-ray absorptiometry (DXA) | 12 weeks
  Body composition will be evaluated by dual energy x-ray absorptiometry at start and end of the study.
Body composition using body composition monitor (BCM) | 12 weeks
  Body composition will be evaluated by bioimpedence analysis using body composition monitor start at and end of the study.

SECONDARY OUTCOMES:
The total score of Short Physical Performance Battery(SPPB) | 12 weeks
  The total score is the sum of 5 times Chair Stand Test(CST) score and balance test score and gait speed test score for 4meter.
The second of 5 times Chair Stand Test | 12 weeks
  Pre test, participants fold their arms across their chest and try to stand up once from a chair. And Measures the time required to perform five rises from a chair to an upright position as fast as possible without the use of the arms.
skeletal muscle mass index(SMI) in cm2/m2 | 12 weeks
  The SMI was calculated according to the following formula: skeletal muscle mass (cm 2) / height 2 (m 2).
Glucose pattern using continuous glucose monitoring system(freestyle libre) | 12 weeks
  Blood glucose is measured using continuous glucose monitoring system(freestyle libre) at start and end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hyon-Seung Yi, Study Chair — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No